CLINICAL TRIAL: NCT02633241
Title: A Pilot Study of Dexmedetomidine-Propofol in Children Undergoing Magnetic Resonance Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph Cravero (Other)
Responsible Party: Sponsor-Investigator, Joseph Cravero, MD, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00019084
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy; Cerebral Palsy; Developmental Delay
Keywords: pediatrics; sedation; dexmedetomidine; propofol; MRI
MeSH Terms: conditions — Epilepsy; Cerebral Palsy; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (bolus and high infusion)-Propofol arm (Other): Patients in this cohort will receive a combination of Dexmedetomidine 1mcg/kg bolus, Dexmedetomidine 1 mcg/kg/hour infusion, and Propofol 100mcg/kg/minute to accomplish an MRI examination.
  Interventions: Drug: Dexmedetomidine bolus and high infusion-Propofol
- Dexmedetomidine (bolus and low infusion)-Propofol arm (Other): Patients in this cohort will receive a combination of Dexmedetomidine 1mcg/kg bolus, Dexmedetomidine 0.5 mcg/kg/hour infusion, and Propofol 100mcg/kg/minute to accomplish an MRI examination.
  Interventions: Drug: Dexmedetomidine bolus and low infusion-Propofol
- Dexmedetomidine (bolus only)-Propofol arm (Other): Patients in this cohort will receive dexmedetomidine 1mcg/kg over 5 minutes and then propofol 2-3mg/kg titrated bolus followed by 100mcg/kg/min infusion to accomplish MRI
  Interventions: Drug: Dexmedetomidine bolus only - Propofol

INTERVENTIONS:
Drug: Dexmedetomidine bolus and high infusion-Propofol — First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1mcg/kg/hour. At the 5 minute point, propofol will be given (2-3mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
  Other Names: Dexmedetomidine-Propofol
  Arms: Dexmedetomidine (bolus and high infusion)-Propofol arm
Drug: Dexmedetomidine bolus and low infusion-Propofol — First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5mcg/kg/hour. At the 5 minute point, propofol will be given (2-3mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
  Other Names: Dexmedetomidine-Propofol
  Arms: Dexmedetomidine (bolus and low infusion)-Propofol arm
Drug: Dexmedetomidine bolus only - Propofol — First, the investigators will begin by administering dexmedetomidine 1mcg/kg over 5 minutes. When this is completed, they will administer propofol 2-3mg/kg titrated bolus followed by 100mcg/kg/min infusion which can also be titrated up or down to a maximum of 300mcg/kg/min to keep the blood pressure and heart rate within 30% of baseline levels.
  Other Names: Dexmedetomidine-Propofol
  Arms: Dexmedetomidine (bolus only)-Propofol arm

SUMMARY:
This is a pilot study to determine if a standard bolus dose and infusion of dexmedetomidine can significantly decrease the dose of propofol (infusion) required for accomplishing an MRI. The investigators studied three arms to examine the effectiveness of dexmedetomidine. Arm 1 was a single bolus of 1.0 mcg/kg with 1.0 mcg/kg/hr infusion followed by propofol infusion. Arm 2 was a bolus of 1.0 mcg/kg with 0.5 mcg/kg/hr infusion followed by propofol infusion. Arm 3 was only a single bolus of 1.0 mcg/kg with no infusion followed by propofol infusion.

DETAILED DESCRIPTION:
A recent publication in the New England Journal of Medicine highlighted the accumulating evidence for neurotoxic effects of anesthetics in animal models and a collection of epidemiologic studies in humans. Recent studies of anesthesia in fetal and neonatal primates are yielding more evidence of neurotoxicity associated with many common anesthesia and sedation techniques (e.g. propofol, etomidate, sevoflurane, desflurane and isoflurane). On the other hand, the data suggests that some alternative sedative agents, such as Dexmedetomidine, may not have the same neurotoxic effect.

Children routinely undergo sedation for MRI scanning with large doses of propofol and other sedatives. Many of these scans occur at young ages when these children may be at risk of neurological injury from sedative exposure. In addition, these scans do not involve any stimulation - which could be protective against neurodegeneration.

The investigators propose a pilot study to determine if a standard bolus dose and infusion of dexmedetomidine can significantly decrease the dose of propofol (infusion) required for accomplishing an MRI. Based on previous work with the combination of propofol with dexmedetomidine for other procedures, the investigators propose a standard dose of dexmedetomidine (1 mcg/kg bolus followed by an infusion at 1.0 mcg/kg/hour, 0.5 mcg/kg/hour, or no infusion). The investigators will augment this sedation with propofol 2-3 mg/kg titrated bolus followed by 100 mcg/kg/min infusion which can also be titrated up or down to a maximum of 300 mcg/kg/min to keep the blood pressure and heart rate within 30% of baseline levels).

The investigators hypothesize that the use of low dose propofol with dexmedetomidine will be effective undergoing MRI while sparing exposure to the high dose of the sedative.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting as out-patients, scheduled to receive an anesthetic for MRI of body (spine, chest, abdomen, and/or pelvis) and/or extremity (arm and/or leg).
2. The subject must be a candidate for the sedation technique described in this study with a natural airway (see exclusion criteria described below). This decision will be made by a staff member of the Department of Anesthesiology.
3. The subjects must be 1 and 12 years.
4. The subject's legally authorized representative has given written informed consent to participate in the study.
5. American Society of Anesthesiologist status I, II, or III

Exclusion Criteria:

1. The subject is residing in the Pediatric Intensive Care Unit, the Cardiac Intensive Care Unit, or Neonatal Intensive Care Unit.
2. Diagnosis of a difficult airway or severe obstructive sleep apnea that is not compatible with spontaneous ventilation in a supine position.
3. Congenital heart disease or history of dysrhythmia.
4. Patient taking digoxin or beta-blocker
5. Anxiolytic medication is ordered before the MRI (e.g., midazolam or ketamine).
6. The subject has a history or a family (parent or sibling) history of malignant hyperthermia.
7. The subject is allergic to or has a contraindication to propofol or dexmedetomidine.
8. The subject has previously been treated under this protocol.
9. The subject has a tracheostomy or other mechanical airway device.
10. The subject has received within the past 12 hours an oral or intravenous alpha-adrenergic, beta-adrenergic agonist, or antagonist drugs (e.g., clonidine, propranolol, albuterol).
11. The subject is not scheduled to receive anesthesia-sedation care for the MRI.
12. The subject received one of the anesthetic regimens for the same MRI during the past six months.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cravero, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rappaport BA, Suresh S, Hertz S, Evers AS, Orser BA. Anesthetic neurotoxicity--clinical implications of animal models. N Engl J Med. 2015 Feb 26;372(9):796-7. doi: 10.1056/NEJMp1414786. PMID 25714157
- [Background] Wu J, Mahmoud M, Schmitt M, Hossain M, Kurth D. Comparison of propofol and dexmedetomedine techniques in children undergoing magnetic resonance imaging. Paediatr Anaesth. 2014 Aug;24(8):813-8. doi: 10.1111/pan.12408. Epub 2014 May 12. PMID 24814202
- [Background] Heard CM, Joshi P, Johnson K. Dexmedetomidine for pediatric MRI sedation: a review of a series of cases. Paediatr Anaesth. 2007 Sep;17(9):888-92. doi: 10.1111/j.1460-9592.2007.02272.x. PMID 17683409
- [Background] Triltsch AE, Welte M, von Homeyer P, Grosse J, Genahr A, Moshirzadeh M, Sidiropoulos A, Konertz W, Kox WJ, Spies CD. Bispectral index-guided sedation with dexmedetomidine in intensive care: a prospective, randomized, double blind, placebo-controlled phase II study. Crit Care Med. 2002 May;30(5):1007-14. doi: 10.1097/00003246-200205000-00009. PMID 12006795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 3.2.2017 and the final patient was enrolled 9.6.2022. Recruitment occurred after mail and phone contact approximately 2 weeks before the study and consent was obtained on the day of the study.
Groups:
- Dexmedetomidine (High)-Propofol Arm: The investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes.
- Dexmedetomidine (Low)-Propofol Arm: The investigators will administer dexmedetomidine 1 mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5 mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100 mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2 mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
- Dexmedetomidine (Bolus Only)-Propofol Arm: The investigators will administer dexmedetomidine 1 mcg/kg over 5 minutes. At the 5 minute point, propofol will be given (2 mg/kg bolus followed by 100 mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2 mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
Period: Overall Study
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Started | 15 | 15 | 41
Completed | 13 | 14 | 28
Not Completed | 2 | 1 | 13

BASELINE CHARACTERISTICS:
Population: The 1st, 2nd, and 3rd arms of this study have been completed and are shown here.
Groups:
- Dexmedetomidine (High)-Propofol Arm: The investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm | Total
Number analyzed (Participants) | 13 | 14 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants] — Population: 71 participants were enrolled but only 55 completed the study. Analysis was only performed on these 55 participants.
  Participants
    <=18 years | 13 | 14 | 28 | 55
    Between 18 and 65 years | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: 71 participants were enrolled but only 55 completed the study. Analysis was only performed on these 55 participants.
  years | 2.6 [1.17 to 5.61] | 4.6 [1.95 to 9.90] | 3.6 [1.56 to 11.87] | 3.6 [1.17 to 11.87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 71 participants were enrolled but only 55 completed the study. Analysis was only performed on these 55 participants.
  Participants
    Female | 3 | 4 | 12 | 19
    Male | 10 | 10 | 16 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 71 participants were enrolled but only 55 completed the study. Analysis was only performed on these 55 participants.
  participants
    United States | 13 | 14 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Dosage/Consumption
Description: Dosage and consumption of dexmedetomidine infusion
Time Frame: Prior to beginning the MRI and throughout the MRI scan - approximately one hour.
Population: Patients who completed the study and received a dexmedetomidine infusion
Measure: Mean (95% Confidence Interval); unit: mcg/kg/min
Groups:
- Dexmedetomidine (High)-Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
- Dexmedetomidine (Low)-Propofol Arm: First, the investigators will administer dexmedetomidine 1 mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5 mcg/kg/hour. At the 5 minute point, propofol will be given (2 mg/kg bolus followed by 100 mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2 mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm
Number analyzed (Participants) | 13 | 14
mcg/kg/min | 0.36 [0.22 to 0.51] | 0.25 [0.17 to 0.33]

2. Primary Outcome: Incidence of Patient Movement and MRI Interruption
Description: If patient moved during their MRI and caused an interruption of the scan.
Time Frame: During the MRI scan, until completion, approximately one hour.
Measure: Number; unit: patients
Groups:
- Dexmedetomidine (High)-Propofol Arm: First, the investigators will administer dexmedetomidine 1.0mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1 mcg/kg/hour. At the 5 minute point, propofol will be given (2 mg/kg bolus followed by 100 mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
- Dexmedetomidine (Low)-Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
- Dexmedetomidine (Bolus Only)-Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Number analyzed (Participants) | 13 | 14 | 28
patients | 2 | 3 | 2

3. Primary Outcome: Incidence of Adverse Events
Description: arterial desaturation, airway obstruction, hypotension and bradycardia
Time Frame: From the time the medication is initiated just (5 minutes) prior to the MRI scan and during the MRI scan and immediately during recovery - approximately one hour and twenty minutes in total.
Measure: Number (95% Confidence Interval); unit: incidents
Groups:
- Dexmedetomidine (High)-Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
- Dexmedetomidine (Low)-Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5 mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Number analyzed (Participants) | 13 | 14 | 28
incidents | 1 [0 to 1] | 1 [0 to 1] | 3 [0 to 3]

4. Primary Outcome: Case Times
Description: Number of minutes from the start of sedation medication administration to the time the patient is adequately sedated for the MRI scan,
Time Frame: Timeframe immediately before the MRI scan while sedation medication is administered - approximately 10 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Dexmedetomidine (Low) -Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5 mcg/kg/hour. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low) -Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Number analyzed (Participants) | 13 | 14 | 28
minutes | 7 [5.5 to 10] | 7 [5.5 to 10] | 7 [5.5 to 10]

5. Secondary Outcome: Incidence of Technique Failure
Description: lack of adequate sedation for MRI scan in spite of the sedation as described above
Time Frame: During the MRI scan until completion - approximately one hour
Measure: Number; unit: incidents
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Number analyzed (Participants) | 13 | 14 | 28
incidents | 0 | 0 | 0

6. Secondary Outcome: Sedation Infusion Time
Description: The number of minutes that the patient was receiving dexmedetomidine infusion
Time Frame: For the duration of the MRI scan - approximately one hour
Population: Patients who completed the study and received a dexmedetomidine infusion
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Dexmedetomidine (High)-Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1.0 mcg/kg/hour. At the 5 minute point, propofol will be given (2 mg/kg bolus followed by 100 mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose of Dexmedetomidine will not be changed. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm
Number analyzed (Participants) | 13 | 14
minutes | 43 [37 to 55] | 50 [31 to 56]

7. Secondary Outcome: Case Duration
Description: total number of minutes in the MRI scanner,
Time Frame: Duration of the MRI scan - approximately one hour
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Dexmedetomidine (High)-Propofol Arm: The investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 1mcg/kg/hour. At the 5 minutes, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine if the child is in an adequate state to begin the MRI scan. If the child is not sufficiently sedated within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
- Dexmedetomidine (Low)-Propofol Arm: The investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5 mcg/kg/hour. At the 5 minutes, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine if the child is in an adequate state to begin the MRI scan. If the child is not sufficiently sedated within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
- Dexmedetomidine (Bolus Only)-Propofol Arm: The investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. At the 5 minutes, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine if the child is in an adequate state to begin the MRI scan. If the child is not sufficiently sedated within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Number analyzed (Participants) | 13 | 14 | 28
minutes | 52.8 (21.2) | 53.3 (16.8) | 40.1 (17.4)

8. Secondary Outcome: Recovery Time
Description: number of minutes in the recovery area until the patient appeared awake (eye opening),
Time Frame: from completion of the MRI scan until prepared for discharge - approximately 90 minutes
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Dexmedetomidine (Low) -Propofol Arm: The investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. Next, the investigators will begin an infusion at 0.5 mcg/kg/hour. At the 5 minutes, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine if the child is in an adequate state to begin the MRI scan. If the child is not sufficiently sedated within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure and sedation will continue at the discretion of the anesthesiologist.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low) -Propofol Arm | Dexmedetomidine (Bolus Only)-Propofol Arm
Number analyzed (Participants) | 13 | 14 | 28
minutes | 63.5 (22) | 60.9 (23.6) | 42.5 (22.4)

ADVERSE EVENTS:
Time Frame: During the MRI scan and recovery - then for one week after the date of discharge.
Description: Enrollment has been completed for all three arms of this study. There are no adverse events to report.
Groups:
- Dexmedetomidine (Bolus Only) -Propofol Arm: First, the investigators will administer dexmedetomidine 1mcg/kg over 5 minutes. At the 5 minute point, propofol will be given (2mg/kg bolus followed by 100mcg/kg/min infusion). The attending clinician will determine whether or not the child is in an adequate state to begin the MRI scan. If the sedative effect of the dexmedetomidine-propofol does not produce a sufficiently sedated state within 10 minutes, a repeat bolus of propofol 2mg/kg will be administered. The dose will be repeated if the child is not adequately sedated in 2 more minutes. At this time infusion rate of propofol will be increased to 200 mcg/kg/minute. If the child is not sedated in 5 more minutes, the outcome will be recorded as a technique failure.
Arm/Group | Dexmedetomidine (High)-Propofol Arm | Dexmedetomidine (Low)-Propofol Arm | Dexmedetomidine (Bolus Only) -Propofol Arm
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/28
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT02633241/Prot_SAP_001.pdf